CLINICAL TRIAL: NCT02516800
Title: Prevalence and Significance of Mutations in Genes Encoding NaPi-co-transporters in the Development of CAVD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: AV-SLC-2014-01
Record Dates: First submitted 2015-02-02; First posted 2015-08-06 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Aortic Valve Calcification; Aortic Stenosis
MeSH Terms: conditions — Aortic Valve, Calcification of; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Full blood Aortic Valve
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Aortic valve calcification: Patients with calcific aortic valve disease, age = 65 years or below
- Control group: Matched control group

SUMMARY:
Mutations in the SLC34A2 gene, that encodes the sodium phosphate co-transporter (NaPi-IIb), cause defect cell-uptake of phosphate, which leads to formation of calcium-phosphate concretions in the lungs as seen in Pulmonary Alveolar Microlithiasis (PAM). Extra pulmonary calcifications, including heart valve calcification, have previously been reported in patients with PAM.

Calcific Aortic Valve Disease (CAVD) is a common disease in the elderly and is characterised by thickening and calcification of the aortic valve leaflets in the absence of rheumatic heart disease. CAVD is present in more than 25% of patients older than age 65 years and is associated with an increased risk of cardiovascular events. Currently, there is no effective therapy for the disease other than surgical aortic valve replacement. Both calcium and phosphate are the major components of calcific deposits in PAM and CAVD. Based on these preliminary findings, the investigators hypothesize that mutations in sodium phosphate co-transporters may play a role in both pulmonary and extra pulmonary calcifications.

Two studies will be performed: 1. A retrospective cross-sectional study including patients with an age ≤ 65 years with CAVD from Denmark and Örebro, will be carried out. Genetic association analysis will be performed to investigate the incidence of common variants in five genes representing sodium phosphate co-transporters (SLC34A1, SLC34A2, SLC34A3, SLC20A1, SLC20A2) compared to healthy controls. Associated genes will subsequently be sequenced to identify possible causal mutations. 2. In a prospective study, aortic valve tissue will be collected from patients with AS undergoing surgical valve replacement. Molecular characterisation of the transporters will be conducted by determining the level of specific mRNA and protein by RT-PCR/qPCR, and Western Blotting, respectively. The localisation and visualisation will be investigated by immunostaining and confocal laser microscopy. Fibroblasts and endothelial cells will be isolated and grown in cultures with subsequent functional studies of the phosphate uptake.

ELIGIBILITY:
Inclusion Criteria:

* Aortic valve calcification
* Informed consent before study participation
* Age: ≥ 18 years ≤ 65 years

Exclusion Criteria:

* Lacking ability to give informed consent
* Radiotherapy towards the thorax
* Severe kidney disease (in dialysis)

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with premature aortic valve stenosis in Denmark and Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2014-05; Primary Completion 2018-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Frequencies of single-nucleotide polymorphisms in genes encoding NaPi co-transporters | Association analyses will be performed after 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Simonsen, Professor, Study Chair — Department of Biomedicine, Aarhus University
Locations (1):
- Department of Biomedicine, Aarhus University, Aarhus, Denmark